CLINICAL TRIAL: NCT04610099
Title: Creating a Laparoscopic Banded Sleeve Gastrectomy
Acronym: RING
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL70754.091.19
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard SG (Active Comparator): 100 patients undergo a standard sleeve gastrectomy
  Interventions: Device: Standard SG
- Banded SG (Experimental): 100 patients undergo a banded sleeve gastrectomy
  Interventions: Device: Banded Sleeve Gastrectomy

INTERVENTIONS:
Device: Banded Sleeve Gastrectomy — banded sleeve gastrectomy
  Other Names: BSG
  Arms: Banded SG
Device: Standard SG — Standard SG
  Arms: Standard SG

SUMMARY:
A Sleeve Gastrectomy (SG) is on the long term not always successful in every patient because weight regain can occur. An intervention to prevent weight regain in the future is to place a silicone band (non-adjustable) around the sleeve (Banded-Sleeve Gastrectomy: BSG) which increases weight loss and decreases weight regain on the longer term. The question is whether primary application of a banded sleeve gives a greater weight loss and / or prevent weight regain in the future versus a standard sleeve gastrectomy.

DETAILED DESCRIPTION:
A Sleeve Gastrectomy (SG) is on the long term not always successful in every patient because weight regain can occur. An intervention to prevent weight regain in the future is to place a silicone band (non-adjustable) around the sleeve (Banded-Sleeve Gastrectomy: BSG) which increases weight loss and decreases weight regain on the longer term. The question is whether primary application of a banded sleeve gives a greater weight loss and / or prevent weight regain in the future versus a standard sleeve gastrectomy.

Study is a prospective, randomized, multi centre trial.

Study population: patients who qualify for a SG are eligible to participate. The primary SG patients may participate if there is a BMI of 35 kg / m2 with a morbidly obesity-related comorbidity or a BMI of 40kg / m2 or higher.

Intervention: The standard SG is compared with a banded-SG (BSG)

ELIGIBILITY:
Inclusion Criteria:

* Alle patients who are eligible for a primary SG

Exclusion Criteria:

* Bariatric surgery in medical history
* BMI > 60kg/m2 or a planned two-stage procedure.
* Patients with a language barrier which may affect the compliance with medical advice
* Patients with a disease not related to morbid obesity, such as Cushing or drug related.
* Chronic bowel disease for example Crohn's disease or colitis Colitis.
* Renal impairment (MDRD <30) or hepatic dysfunction (liver function twice the normal values)
* Pregnancy during follow-up
* Patients with treatment-resistant reflux symptoms. Defined as reflux persistent symptoms despite the use of a minimum dose of proton-pump inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Total Body Weight loss (%TBWL) | 3 years
  ((preoperative weight - current weight) / (preoperative weight)) x 100%. Weight loss measured in kilograms

SECONDARY OUTCOMES:
Percentage Excess Weight Loss (%EWL) | 3 years
  ((Preoperative weight - current weight) / (preoperative weight - ideal weight at BMI 25)) x 100%. Weight loss measured in kilograms
Quality of life due to questionnaire | 3 years
  Measuring BAROS
Quality of life due to questionnaire | 3 years
  BODY-Q: Patient reporterd outcome measurement, The questionnaire measures three domains; health related quality of life, appearance and experience of healthcare. Each domain is composed of independently functioning scales. Each scale contains different statements, which can be scored on four levels ranging from totally disagree to totally agree or from never to always. The sum of levels ranging from 1 to 4 is the raw score of the different scales. This score can be converted into a Rasch Transformed score ranging from 0, worst score, to 100, best score.
Quality of life due to questionnaire | 3 years
  SF-36; consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Gastroesophageal reflux disease | 3 years
  Measuring GERD-HRQL questionnaire, a higher score on the questionnaire indicates more complaints of gastroesophageal reflux disease.
Reduction of comorbidities | 3 years
  Measuring reduction of diabetes, hypertension, dyslipidemia, osteoarticular disease, OSA

CONTACTS AND LOCATIONS:
Overall Officials: Hazebroek, Principal Investigator — Rijnstate Hospital
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Zuyderland Medisch Centrum, Heerlen, Limburg
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided